CLINICAL TRIAL: NCT06675175
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Study to Assess the Safety, Tolerability, and Pharmacodynamics of AZD4144 in Participants With Established Atherosclerotic Cardiovascular and Chronic Kidney Disease
Brief Title: A Phase 1b Study to Assess the Safety, Tolerability, and Pharmacodynamics of AZD4144 in Participants With Established Atherosclerotic Cardiovascular and Chronic Kidney Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9441C00001; 2024-516840-24-00 (Registry Identifier: EU-CT Number)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease; Atherosclerotic Cardiovascular Disease
Keywords: Cardiorenal disease; Estimated glomerular filtration rate; Nucleotide-binding domain, leucine-rich-containing family, pyrin domain-containing-3 (NLRP3) cryopyrin; inflammatory cytokines
MeSH Terms: conditions — Renal Insufficiency, Chronic; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4144 (Experimental): Participants will receive oral dose of AZD4144 for 28 days.
  Interventions: Drug: AZD4144
- Placebo (Placebo Comparator): Participants will receive oral dose of Placebo for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD4144 — Oral solution of AZD4144 will be given to randomised participants as per the arm they have been assigned.
  Arms: AZD4144
Other: Placebo — Placebo will be given orally to randomized participants as per the arm they are assigned.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and the pharmacodynamics (PD) of AZD4144 following oral administration in participants with atherosclerotic cardiovascular disease (ASCVD) and chronic kidney disease (CKD).

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, double blind, placebo-controlled study and will be conducted in participants with established ASCVD and CKD with persistent inflammation (High-sensitivity C-reactive protein [hsCRP] > 2 mg/L and eGlomerular filtration rate [eGFR] ≥ 30 to < 60 mL/min/1.73m2). The participants will be randomized in the 1:1 ratio to either receive treatment with AZD4144 or placebo.

The study will be comprised of:

* A screening period of 28 days
* Treatment period where each participant will either receive oral dose of AZD4144 or placebo for 28 days.
* A follow-up visit (Day 35 ±1) and a Final Follow-up (on Day 56±1) post first dose administration.

The total duration of the study will be approximately 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with established ASCVD history of one or more of the following

  1. Prior Myocardial infarction (MI) (>60 days from index event) or coronary revascularization procedure like coronary stenting or Coronary artery bypass graft (CABG)
  2. Prior ischemic stroke (>60 days from index event)
  3. Symptomatic Peripheral Arterial Disease
* Chronic kidney disease defined as eGlomular filtration rate (eGFR) ≥ 30 to < 60 mL/min/1.73 m2
* Serum hsCRP > 2 mg/L
* Body mass index ≥ 18 to ≤ 45 kg/m2
* All females must have a negative pregnancy test at the Screening Visit and at the randomization visit

  1. Sexually active male participants with partner of childbearing potential must adhere to the contraception methods
  2. Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception
  3. Females of non-childbearing potential must be confirmed at the Screening visit

Key Exclusion Criteria:

* History of malignancy within the last 5 years
* History of MI, coronary revascularization, stroke or revascularization for peripheral arterial disease in the 60 days prior to Screening
* Active systemic infection within 30 days
* Clinically significant active and chronic infections within 60 days prior to randomization
* Clinically significant recurrent infection (≥ 2× during the last 12-month period).
* Renal transplant participants, participants on dialysis, and those with a history of acute kidney injury in the past 12 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From first dose (Day 1) until Follow-up (Day 56±1)
  The safety and the tolerability of AZD4144 compared with placebo will be evaluated.
Relative change from baseline to 4 weeks in systemic Interleukin-6 (IL-6) levels | Day 1 to Day 28
  The effect of AZD4144 on circulating inflammatory biomarker IL-6 compared with placebo will be evaluated.

SECONDARY OUTCOMES:
Relative change from baseline to 4 weeks in systemic IL-18 and High-sensitivity C-reactive protein (hsCRP) levels | Day 1 to Day 28
  The effect of AZD4144 on circulating inflammatory biomarkers IL-18 and hsCRP compared with placebo will be evaluated.
Maximum plasma drug concentration (Cmax) | Day 1 to Day 28 (pre-dose), Day 1 and Day 22±1 (post-dose)
  The Cmax after administration of AZD4144 in participants with ASCVD and CKD will be evaluated.
Time to reach maximum observed concentration (tmax) | Day 1 to Day 28 (pre-dose), Day 1 and Day 22±1 (post-dose)
  The tmax after administration of AZD4144 in participants with ASCVD and CKD will be evaluated.
Observed lowest concentration before the next dose is administered (Ctrough) | Day 1 to Day 28 (pre-dose), Day 1 and Day 22±1 (post-dose)
  The Ctrough after administration of AZD4144 in participants with ASCVD and CKD will be evaluated.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (9):
  - Research Site, Glendale, California
  - Research Site, Daytona Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tampa, Florida
  - Research Site, Farmington Hills, Michigan
  - Research Site, The Bronx, New York
  - Research Site, Sherman, Texas
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sofia
- Hungary (2):
  - Research Site, Gyöngyös
  - Research Site, Kistarcsa
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/